CLINICAL TRIAL: NCT01017094
Title: Can Silversulfadiazine Prevent Pin-site Infection in Open Tibial Fracture?: A Randomized Controlled Trial
Brief Title: Pin Site Infection Prevention for Open Tibial Fracture
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Secretariate,Department of Orthopaedic Surgery, Faculty of Medicine, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC 50/369-006
Record Dates: First submitted 2009-11-17; First posted 2009-11-20 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Tibial Fracture
Keywords: Pin-site infection; silversulfadiazine; open fracture; open tibial fracture underwent external fixator
MeSH Terms: conditions — Tibial Fractures; Fractures, Open

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- dry dressing (Experimental): local application
  Interventions: Drug: silversulfadiazine

INTERVENTIONS:
Drug: silversulfadiazine — apply once a day

SUMMARY:
This study aimed to compare the efficacy of pin-tract infection prevention between silversulfadiazine and dry dressing.

Methods: 30 patients with an open tibial fracture admitted to Songklanagarind hospital from September 2007 to June 2008 and treated by emergency debridement and external fixation were randomized into two groups, one treated with silversulfadiazine for infection prophylaxis (15) and a control group treated with dry dressing only (15). All patients were followed until the external fixator was removed. Pin-site infections were assessed and graded at each follow-up visit by an orthopaedist blinded to the mode of treatment. A culture from the pin site was done if an infection occurred.

ELIGIBILITY:
Inclusion Criteria:

* Open tibial fracture treated with external fixator age between 15-60 years

Exclusion Criteria:

* Immunocompromised patients (diabetes, HIV or malignancy)

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
incidence of pin site infection | 2 years

SECONDARY OUTCOMES:
type of organism | 2 years
severity of pin site infection | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Boonsin Tangtrakulwanich, MD.,Ph.D, Principal Investigator — Faculty of Medicine, Prince of Songkla University
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand